CLINICAL TRIAL: NCT01919671
Title: A Randomized, Double-blind, Placebo Controlled Evaluation, Multicenter Clinical Study of Tongxinluo Capsule in Ischemic Stroke Patients
Brief Title: Tongxinluo Capsule in Ischemic Stroke Patients（TISS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: yongjun wang (Other Government)
Responsible Party: Sponsor-Investigator, yongjun wang, Vice president of Beijing Tiantan Hospital, Ministry of Science and Technology of the People´s Republic of China
Organization: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: yl-yxb09-lcsyfa-201301
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; Tongxinluo capsule
MeSH Terms: conditions — Ischemic Stroke | interventions — tongxinluo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tongxinluo capsule (Experimental): Tongxinluo capsule,4 granules,t.i.d. po,for 90 days
  Interventions: Drug: Tongxinluo capsule
- placebo capsule (Placebo Comparator): placebo capsule,4 granules,t.i.d. po,for 90 days
  Interventions: Drug: placebo capsule

INTERVENTIONS:
Drug: Tongxinluo capsule — for 90 days
  Other Names: Yiling Pharmaceutical，Z19980015
  Arms: Tongxinluo capsule
Drug: placebo capsule — for 90 days
  Other Names: placebo
  Arms: placebo capsule

SUMMARY:
The purpose of this study is to assess the effects in improving life self-care ability of stroke patients after taking Tongxinluo Capsule(within 72 hours after onset) versus Placebos for 90 days.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, placebo controlled, multi-center trial. We aim to enroll a total of 1968 individuals(984 cases in each group) with acute ischemic stroke less than 72 hours after onset. Participants will be randomized into Tongxinluo capsule treatment group with the capsule administration of 4 granules tid. for 90 days, while the patients in the control group receive placebo capsule. NIH Stroke Score of the subjects is 4-22 at randomization. Evaluations of efficacy and safety will be taken at baseline, 7 days, discharge date and 90 days. Neuroimaging [magnetic resonance imaging (MRI) scans] will be obtained at baseline and 90 days after therapy. The primary efficacy endpoint is the proportion of Modified Rankin Scale (mRS) ≤1 at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stoke within 72 after onset, confirmed by MRI or CT.
* Age 35-75 years, inclusive.
* Patients with the first attack or patients with stroke history(modified Rankin Scale score 0-1).
* Clear signs of localization of nervous system, NIHSS score 4 to 22.
* Patient or proxy has signed informed consent.

Exclusion Criteria:

* Hemorrhage diseases according to head CT or MRI, such as hemorrhagic stroke, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, haemorrhage after cerebral infarction.
* Transient Ischemic Attack (TIA).
* Severe disturbance of consciousness: 1a of NIHSS score>1 point; Difficulty in swallowing, unable to take oral capsules; any of 5a, 5b, 6a, 6b of NIHSS score>2 point.
* Convinced of stroke caused by brain tumor, brain trauma, hemopathy, etc.
* Hemorrhagic tendency patients.
* Patients with endovascular treatment after the onset of stroke.
* Patients with dementia, severe Parkinson's disease, mental disorders, limb dysfunction caused by other diseases or other conditions that may affect the therapeutic efficacy.
* Uncontrolled hypertension (≥200 mmHg systolic or ≥110 mmHg diastolic) or hypotension (≤90 mmHg systolic or ≤60mmHg diastolic); severe hyperglycemia(blood glucose ≥400 mg/dl) or hypoglycemia( blood glucose≤50 mg/dl).
* Severe hepatic insufficiency defined as transaminase values > 2x upper limit of normal; severe renal insufficiency defined as values serum creatinine> 1.5x upper limit of normal; cardiac dysfunction or other serious systemic disease with life expectancy ≤3 months.
* Patients with concurrent malignancy or ongoing anti-tumor therapy.
* Patients with history of being allergic to the trial medicine.
* Pregnancy, breastfeeding or potential pregnancy.
* Within three months or currently participating in another investigational study.
* Any other condition that in the opinion of the investigator should preclude study participation.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2007 (Actual)
Dates: Start 2014-03; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Modified Rankin Scale (mRS) less than or equal to 1 at 90 days. | 90 days

SECONDARY OUTCOMES:
Proportion of patients with National Institutes of Health Stroke Score (NIHSS) reaching 0-1 or reduction 4 points . | Baseline, 7days, discharge date, 90 days
Proportion of patients with Bathel Index（BI）score more than 85. | Baseline, 7days, discharge date, 90 days
Continuous changes of Modified Rankin Scale score. | Baseline, 7days, discharge date, 90 days
Incidence of ischemic cerebrovascular disease (ischemic stroke/TIA/ new ischemic lesion in MRI Images. | 90 days
Incidence of new combination clinical vascular events (ischemic stroke/ hemorrhagic stroke/ TIA/ MI/ vascular death). | 90 days

OTHER OUTCOMES:
MR indicated symptomatic or non-symptomatic cerebral infarction emerging | 90 days
  Compared with baseline MRI, re-examination of MRI shows new infarct diagnosed by DWI or FLARI (including new infarct and enlargement of infarct size) in areas other than the original infarct in DWI and FLAIR-sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, professor, Study Director — Beijing Tiantan Hospital
Locations (1):
- Beijing TianTan Hospital,Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dong Y, Jiang K, Li Z, Zhou Y, Ju B, Min L, He Q, Fan P, Hu W, Qu H, Wu H, Pan C, Cao Y, Lou X, Zhang G, Zhang J, Hu F, Dong Q; TISS Trial Investigators. Tongxinluo and Functional Outcomes Among Patients With Acute Ischemic Stroke: A Randomized Clinical Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2433463. doi: 10.1001/jamanetworkopen.2024.33463. PMID 39325453